CLINICAL TRIAL: NCT07021846
Title: Hypofractionated Radiotherapy With Dose Escalated Concomitant Boost for Breast Cancer: a Phase 2 Trial
Brief Title: Dose Escalated Concomitant Boost Radiotherapy for Early Breast Cancer
Acronym: DEBoRa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63/19 PAR ComEt CBM
Record Dates: First submitted 2025-05-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: tumor bed boost; radiotherapy; hypofractionation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypofractionated arm + concomitant tumor bed boost (Experimental): Hypofractionation arm, 40 Gy in 15 fractions (2.67 Gy per fraction over 3 weeks) and a tumor bed boost to a total dose of 52.5 Gy in 15 fractions (3.5 Gy per fraction over 3 weeks).
  Interventions: Radiation: hypofractionated radiotherapy with tumor bed boost

INTERVENTIONS:
Radiation: hypofractionated radiotherapy with tumor bed boost — hypofractionated radiotherapy with concomitant/simultaneous tumor bed boost

SUMMARY:
The goal of this prospective, single-arm, phase II, non-randomized trial is to evaluate an hypofractionation schedule with high dose simultaneous integrated tumor bed boost in early breast cancer patients.

The main question[s] it aims to answer are:

* evaluate the rate of all grades of radiation-induced fibrosis at 4 years.
* evaluate poor/fair cosmesis rate Participants will be treated with hypofractionated radiotherapy (RT) to whole breast with a dose of 40.05 Gy in 15 fractions (2.67 Gy/die) and a concomitant tumor bed dose of 52.5 Gy (3.5 gy/die)

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase II, non-randomized clinical trial that will test an hypofractionated schedule with high dose simultaneous integrated tumor bed boost set on a previous dose finding study. Patients will be treated with hypofractionated RT to whole breast with a dose of 40.05 Gy in 15 fractions (2.67 Gy/die) and a concomitant tumor bed dose of 52.5 Gy (3.5 gy/die). The study population will include early breast cancer patients with younger age (< or= 50 years) and additional risk factors for local recurrence.

The primary objective of the study is to evaluate the rate of radiation-induced fibrosis at 4 years.The expected enrollment is 132 patients in 6 years. Each patient must have a minimum follow-up of 4 years.

The secondary objective is to evaluate cosmesis; other objectives are to evaluate quality of life (QoL) and the rate of local control.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven breast cancer who have undergone conservative surgery
* at least 3 inserted clips
* age: from 18 years old to 50 years
* at least one of the following risk factors: N1 disease, LVI, extensive intraductal component (>25%), close margins (<4 mm), non-hormone-sensitive disease, grading 3
* ECOG performance status < 2
* adequate bone marrow (haemoglobin concentration > 8 g/dl, white blood cell count > 3000/mm3, platelet count > 75000).

Exclusion Criteria:

* Previous chest radiation treatment
* Bilateral breast cancer
* Neoadjuvant chemotherapy
* BMI > 35
* Collagen diseases
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 132 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Breast fibrosis | baseline, each year up to 4 years after radiotherapy
  Rate of all grades breast fibrosis evaluated by means of Common Terminology Criteria for Adverse Events (CTCAE) v. 5 scale

SECONDARY OUTCOMES:
Breast cosmesis | baseline, each year up to 4 years after radiotherapy
  Rate of fair and poor cosmesis evaluated by means of European Organisation for Research and Treatment of Cancer (EORTC) Cosmetic Rating System for Breast Cancer
Quality of Life (QOL) | baseline, each year up to 4 years after radiotherapy
  Quality of Life evaluated by means of European Organization for Research and Treatment-QOL questionnaire (EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Locations (1):
- Università Campus Biomedico, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartelink H, Horiot JC, Poortmans P, Struikmans H, Van den Bogaert W, Barillot I, Fourquet A, Borger J, Jager J, Hoogenraad W, Collette L, Pierart M; European Organization for Research and Treatment of Cancer Radiotherapy and Breast Cancer Groups. Recurrence rates after treatment of breast cancer with standard radiotherapy with or without additional radiation. N Engl J Med. 2001 Nov 8;345(19):1378-87. doi: 10.1056/NEJMoa010874. PMID 11794170
- [Background] Romestaing P, Lehingue Y, Carrie C, Coquard R, Montbarbon X, Ardiet JM, Mamelle N, Gerard JP. Role of a 10-Gy boost in the conservative treatment of early breast cancer: results of a randomized clinical trial in Lyon, France. J Clin Oncol. 1997 Mar;15(3):963-8. doi: 10.1200/JCO.1997.15.3.963. PMID 9060534
- [Background] Vrieling C, Collette L, Fourquet A, Hoogenraad WJ, Horiot JC, Jager JJ, Pierart M, Poortmans PM, Struikmans H, Van der Hulst M, Van der Schueren E, Bartelink H. The influence of the boost in breast-conserving therapy on cosmetic outcome in the EORTC "boost versus no boost" trial. EORTC Radiotherapy and Breast Cancer Cooperative Groups. European Organization for Research and Treatment of Cancer. Int J Radiat Oncol Biol Phys. 1999 Oct 1;45(3):677-85. doi: 10.1016/s0360-3016(99)00211-4. PMID 10524422
- [Background] Yarnold J, Ashton A, Bliss J, Homewood J, Harper C, Hanson J, Haviland J, Bentzen S, Owen R. Fractionation sensitivity and dose response of late adverse effects in the breast after radiotherapy for early breast cancer: long-term results of a randomised trial. Radiother Oncol. 2005 Apr;75(1):9-17. doi: 10.1016/j.radonc.2005.01.005. Epub 2005 Mar 16. PMID 15878095
- [Background] Ippolito E, Rinaldi CG, Silipigni S, Greco C, Fiore M, Sicilia A, Trodella L, D'Angelillo RM, Ramella S. Hypofractionated radiotherapy with concomitant boost for breast cancer: a dose escalation study. Br J Radiol. 2019 Mar;92(1095):20180169. doi: 10.1259/bjr.20180169. Epub 2018 Nov 28. PMID 30433824